CLINICAL TRIAL: NCT00122564
Title: Phase I Study Evaluating the Systemic and Mucosal Safety and Immunogenicity of a Recombinant HIV-1 Gp 160 (MN/LAI) Administered by Transmucosal (Nasal or Vaginal) Routes, Alone or Formulated With DC-Chol, in HIV Negative Volunteers (ANRS VAC14)
Brief Title: Study of HIV-1 Rgp-160 Administered by Mucosal Routes in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS VAC14
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2005-11-11 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infections
Keywords: HIV Vaccines; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — 3-(N-(N',N'-dimethylaminoethane)carbamoyl)cholesterol

INTERVENTIONS:
Biological: HIV-1 gp 160
Biological: DC-Chol

SUMMARY:
It is probable that a mucosal approach is necessary for a prophylactic HIV vaccine protecting against sexually transmitted infection. Mucosal immune responses have been almost non-existent in trials of HIV vaccine candidates in which the antigen was delivered systemically. This study will test the safety and immune response of a recombinant HIV-1gp160 by nasal and mucosal routes alone or formulated with DC-Chol in healthy volunteers.

DETAILED DESCRIPTION:
It's probable that a mucosal approach is necessary for prophylactic HIV vaccine protecting against sexually transmitted infection. Although mucosal immune responses have been almost non-existent in trials of HIV vaccine candidates in which the antigen was delivered systematically.

Several animal models have also demonstrated the importance or a mucosal IgA response for protection against viral infections. Mucosal S IgA are essential effectors having different mechanisms of action agglutination of pathogens, interaction with cellular receptor, transcytosis of immune complexes, intracellular clearance of virus.

Gp 160 induces the majority of neutralizing Abs activity in patients serum and the immunogenicity of gp 160 can be improved by using and adjuvant such as DC-chol because of its properties to increase the permeation of the nasal epithelium and to facilitate systemic delivery of the vaccine antigen.

Before beginning mucosal vaccine trial, we previously tested and validated procedures to collect and process secretion fluids on 6 HIV-1 infected women (K. Petitprez et al, 4th European mucosal immunology group meeting, Lyon France, 8-10 october 2004).

ELIGIBILITY:
Inclusion Criteria:

* Women chosen in a uniform selection process specifically designed by the ANRS (French National Agency for Research on AIDS and Viral Hepatitis)
* For women of child-bearing age : use of effective contraception
* Normal clinical status
* Ability to accept collection of secretion fluids;
* Ability to sign informed consent

Exclusion Criteria:

* Pregnancy

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36
Dates: Start 2003-06; Study Completion 2005-04

PRIMARY OUTCOMES:
Systemic and mucosal safety evaluated by 3 independent physicians at week 0, 4, 6 and 48 and 2 days after each mucosal administration

SECONDARY OUTCOMES:
Immune response by ELISA for anti-gp 160 IgA or IgG and by functional in vitro assay

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Pialoux, MD, Principal Investigator — Hopital Tenon Paris
Locations (1):
- Hopital Tenon, Paris, France